CLINICAL TRIAL: NCT04165200
Title: Fecal Microbiota Transplantation as a Therapeutic Strategy for Patients Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Dr. Adrian Camacho Ortiz, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IF18-00008
Record Dates: First submitted 2019-11-04; First posted 2019-11-15 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: HIV Infections
Keywords: HIV infection, fecal microbiota transplantation
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Prospective controlled study experimental comparative
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither patients, nor investigators are allowed to know about which group of patients is going to receive placebo and which one faecal microbiota capsules. The laboratory that provide us the capsules is going to divide and randomize our sample of patients, and also register the information in a data base.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving FMT capsules and ART (Active Comparator): 1. ART Start at week 0 non-stop.
  2. FMT. The frozen capsules will be ingested orally at a frequency of 15 capsules every 12 hours for four doses 7 days prior ART start and on weeks 0, 4, 8 and 12 after ART start. Each capsule must be ingested over a period no longer than 1 hour of the anterior capsule.
  3. Blood samples Week 0, 4, 8, 12 and 24. Taken through peripheral vein puncture with the extraction of 10 ml of venous blood to monitor the CD4 lymphocytes count and HIV viral load.
  4. Feces samples from each patient will be taken during medical consultation on week 0, 8 and 24 after ART start to evaluate the modification of the intestinal microbiome.
  5. Medical consultations will be made on days -7 to ART start, day 1, 30, 60, 90 and 120 after ART start, where clinical examination and elimination criteria will be evaluated.
  Interventions: Diagnostic Test: Blood and feces samples
- Patients receiving placebo capsules (Placebo Comparator): 1. ART Start at week 0 non-stop.
  2. Placebo capsules. The frozen capsules will be ingested orally at a frequency of 15 capsules every 12 hours for four doses 7 days prior ART start and on weeks 0, 4, 8 and 12 after ART start. Each capsule must be ingested over a period no longer than 1 hour of the anterior capsule.
  3. Blood samples Week 0, 4, 8, 12 and 24. Taken through peripheral vein puncture with the extraction of 10 ml of venous blood to monitor the CD4 lymphocytes count and HIV viral load.
  4. Feces samples from each patient will be taken during medical consultation on week 0, 8 and 24 after ART start to evaluate the modification of the intestinal microbiome.
  5. Medical consultations will be made on days -7 to ART start, day 1, 30, 60, 90 and 120 after ART start, where clinical examination and elimination criteria will be evaluated.
  Interventions: Diagnostic Test: Blood and feces samples

INTERVENTIONS:
Diagnostic Test: Blood and feces samples — Blood samples are going to be taken by puncturing peripheral vein extraction with 10 ml of venous blood for later biweekly to monitor in person and therefore monitor immune status with biomarkers T lymphocyte subclass CD4 and viral load. A total of four blood samples will be taken at weeks 4, 8, 12 and 24 of recruitment.
  A total of four feces samples are going to be required during the study, to evaluate the changes on the microbiota of the patient. 1 week before the patients start their HAART, the same day the patients initiate their HAART, 8 weeks after they started HAART and 24 weeks after HAART.

SUMMARY:
Patients eligible for the study will be selected on Fridays during the HIV consultation at the Infectious Diseases Department. Patients that meet the inclusion and exclusion criteria, will be randomized and assigned in two groups 1:1. A group will start intervention with FMT (fecal matter transplant) through frozen capsules and after seven days, antiretroviral therapy (ART) will be started. Patients in the other group will be given placebo capsules and after seven days ART will be started. The frozen capsules of FMT will be ingested orally with a frequency of 15 capsules every 12 hours for 4 doses 7 days prior ART start and on weeks 0, 4, 8 and 12 after ART start. Subsequently, blood samples will be taken to monitor the immune status with CD4 T lymphocytes and HIV viral load during week 0, 4, 8, 12 and 24 after ART start.

Throughout the study period, subjects can carry out a free diet, moderate alcohol intake, perform their daily activities and abstain from any of the elimination criteria. Medical consultations will be made on days -7 to ART start, day 1, 30, 60, 90 and 120 after ART start, where clinical examination and elimination criteria will be evaluated.

DETAILED DESCRIPTION:
Study design: Prospective controlled study experimental comparative Study duration: 1 year The number of patients to enroll: 20 patients. After being randomized, selected patients who meet the criteria for inclusion and exclusion will be assigned 1:1 in two groups. A group will start treatment with FMT through frozen capsules, and ART at the same time; and another group will star placebo capsules and ART.

The frozen capsules will be ingested orally at a frequency of 15 capsules every 12 hours for four doses 7 days prior ART start and on weeks 0, 4, 8 and 12 after ART start. Each capsule must be ingested over a period no longer than 1 hour of the anterior capsule.

Subsequently, blood samples will be taken through peripheral vein puncture with the extraction of 10 ml of venous blood to monitor the immune status with CD4 T lymphocytes and HIV viral load. A total of 4 blood samples will be taken during week 4, 8, 12 and 24 after ART start.

Medical consultations will be made every 4 weeks, on days -7 days prior ART start, day 1, 30, 60, 90 and 120 where vital signs, symptoms or signs of organ systems, determination of weight, BMI, adverse effects and elimination criteria will be assessed.

In addition, feces samples from each patient will be taken during medical consultation on week 0, 8 and 24 after ART start to evaluate the modification of the intestinal microbiome after the intervention on both groups.

During the study period, subjects may carry a free diet, moderate intake of alcohol and perform their daily activities as they refrain free from any of the elimination criteria.

The study will last 1 year and the samples taken will be frozen and stored in the Infectious Diseases Department of the Hospital.

Selection of Fecal Microbiota donors:

The selection of fecal microbiota donors is based on:

* Medical history, body weight, no medication uses such as antibiotics and proton pump inhibitors, no trips and no diarrhea 6 months prior donation.
* The absence of chronic infections such as Hepatitis B, Hepatitis C, and HIV determined by immunoassay.
* Negative Rose Bengal test and V.D.R.L
* Normal complete blood count and liver function tests.

Fecal sample analysis:

1. Fresh microscopy analysis to detect leukocytes and parasites (including protozoa and helminths)
2. Stool culture to rule out the presence of enteropathogens, including Salmonella spp., Shigella spp., Aeromonas spp., Plesiomonas spp., Vibrio spp. and Clostridiodes diffcile.
3. Gastrointestinal panel by multiple polymerase chain reaction (PCR) using BioFire Filmarray which includes the detection of:

   Bacteria: Campylobacter (C. jejuni, C. coi, C. upsaliensis), Clostridiodes difficile (toxins A / B), Plesiomonas shigelloides, Salmonella spp., Yersinia enterocolitica, Vibrio (V. parahaemolytic , V. vulnificus and V. cholerae), Escherichia coli O157: H7, enteroaggregative E. coli (EAEC), enteropathogenic E. coli (EPEC), enterotoxigenic E. coli (ETEC), Shiga toxin producing E. coli (STEC) stx1 / stx2, Shigella sp. enteroinvasive E. coli (EIEC).

   Virus: Adenovirus F 40/41, Astrovirus, Norovirus GI / GII, Rotavirus A, Sapovirus (I, II, IV and V) Parasites: Cryptosporidium sp., Cyclospora cayetanensis, Entamoeba histolytica and Giardia lamblia.
4. Detection of genes associated with drug resistance by endpoint PCR; including genes encoding extended spectrum beta-lactamases (TEM, CTX; SHV, CMY) and carbapenemases (VIM, NDM, IMP, KPC, OXA-48).

Once all the stages of evaluation are completed only negative subjects for all the tests and in which there is no evidence of infection are selected as donors. The scrutiny and laboratory tests are considered valid during the following 4 weeks, so if new donation of feces is required, the process will be carried out again.

Sample Preparation fecal microbiota All samples will be mixed with 10% glycerol and frozen at -70°C in a period not exceeding 60 minutes after collection. They will be mixed and then suspended in saline 0.9%. The final mixture will be filtered to remove particles greater than 330 microns, finally adding glycerol as cryoprotectant. This mixture is carried to the encapsulation process using sterile capsules for enteral liberation, in two sizes. The first capsule is filled with a mixture of feces and sealed with its counterpart, and then the sealed capsule becomes encapsulated in a second capsule. The final product is stored frozen until 60 minutes before use. The administration will only be oral.

ELIGIBILITY:
Inclusion criteria:

* Patients over 18 years
* Confirmed HIV infection with any CD4 lymphocyte count
* Patients at the beginning of the study only taking antibiotic prophylaxis according to the CD4 lymphocyte count
* Patients agree to participate in the study through a signed informed consent

Exclusion criteria:

* Patients receiving probiotics
* Patients with anatomical abnormalities of the digestive tract such as colostomy or ileostomy
* Patients with previous bowel resection
* Patients with impaired AST and / or ALT greater than 4 times its normal value
* Hemodialysis patients Patients with gastrointestinal bleeding in the last 12 weeks
* Patients undergoing colonoscopy in the last 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Levels of CD4 cells | 6 months
  The efficacy of FMT in obtaining a faster immunologic response measured in rise of CD4 lymphocyte countTMF capsules, will have a faster rise in cell count than those who don´t receive them.

SECONDARY OUTCOMES:
Tolerability of FMT capsules | 6 months
  Number of Participants with FMT related Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Arts EJ, Hazuda DJ. HIV-1 antiretroviral drug therapy. Cold Spring Harb Perspect Med. 2012 Apr;2(4):a007161. doi: 10.1101/cshperspect.a007161. PMID 22474613
- [Background] Zulfiqar HF, Javed A, Sumbal, Afroze B, Ali Q, Akbar K, Nadeem T, Rana MA, Nazar ZA, Nasir IA, Husnain T. HIV Diagnosis and Treatment through Advanced Technologies. Front Public Health. 2017 Mar 7;5:32. doi: 10.3389/fpubh.2017.00032. eCollection 2017. PMID 28326304
- [Background] Brenchley JM, Paiardini M, Knox KS, Asher AI, Cervasi B, Asher TE, Scheinberg P, Price DA, Hage CA, Kholi LM, Khoruts A, Frank I, Else J, Schacker T, Silvestri G, Douek DC. Differential Th17 CD4 T-cell depletion in pathogenic and nonpathogenic lentiviral infections. Blood. 2008 Oct 1;112(7):2826-35. doi: 10.1182/blood-2008-05-159301. Epub 2008 Jul 29. PMID 18664624
- [Background] Mutlu EA, Keshavarzian A, Losurdo J, Swanson G, Siewe B, Forsyth C, French A, Demarais P, Sun Y, Koenig L, Cox S, Engen P, Chakradeo P, Abbasi R, Gorenz A, Burns C, Landay A. A compositional look at the human gastrointestinal microbiome and immune activation parameters in HIV infected subjects. PLoS Pathog. 2014 Feb 20;10(2):e1003829. doi: 10.1371/journal.ppat.1003829. eCollection 2014 Feb. PMID 24586144
- [Background] Dillon SM, Lee EJ, Kotter CV, Austin GL, Dong Z, Hecht DK, Gianella S, Siewe B, Smith DM, Landay AL, Robertson CE, Frank DN, Wilson CC. An altered intestinal mucosal microbiome in HIV-1 infection is associated with mucosal and systemic immune activation and endotoxemia. Mucosal Immunol. 2014 Jul;7(4):983-94. doi: 10.1038/mi.2013.116. Epub 2014 Jan 8. PMID 24399150
- [Background] Hunt PW. Th17, gut, and HIV: therapeutic implications. Curr Opin HIV AIDS. 2010 Mar;5(2):189-93. doi: 10.1097/COH.0b013e32833647d9. PMID 20543599
- [Background] Samji H, Cescon A, Hogg RS, Modur SP, Althoff KN, Buchacz K, Burchell AN, Cohen M, Gebo KA, Gill MJ, Justice A, Kirk G, Klein MB, Korthuis PT, Martin J, Napravnik S, Rourke SB, Sterling TR, Silverberg MJ, Deeks S, Jacobson LP, Bosch RJ, Kitahata MM, Goedert JJ, Moore R, Gange SJ; North American AIDS Cohort Collaboration on Research and Design (NA-ACCORD) of IeDEA. Closing the gap: increases in life expectancy among treated HIV-positive individuals in the United States and Canada. PLoS One. 2013 Dec 18;8(12):e81355. doi: 10.1371/journal.pone.0081355. eCollection 2013. PMID 24367482
- [Background] Bandera A, De Benedetto I, Bozzi G, Gori A. Altered gut microbiome composition in HIV infection: causes, effects and potential intervention. Curr Opin HIV AIDS. 2018 Jan;13(1):73-80. doi: 10.1097/COH.0000000000000429. PMID 29045252
- [Background] Desai SN, Landay AL. HIV and aging: role of the microbiome. Curr Opin HIV AIDS. 2018 Jan;13(1):22-27. doi: 10.1097/COH.0000000000000433. PMID 29035948
- [Background] Lozupone CA, Li M, Campbell TB, Flores SC, Linderman D, Gebert MJ, Knight R, Fontenot AP, Palmer BE. Alterations in the gut microbiota associated with HIV-1 infection. Cell Host Microbe. 2013 Sep 11;14(3):329-39. doi: 10.1016/j.chom.2013.08.006. PMID 24034618